CLINICAL TRIAL: NCT07014722
Title: Contact Activation of Coagulation in Newly Inserted Central Catheters - a Randomized Controlled Trial
Brief Title: Contact Activation of Coagulation in Newly Inserted Central Venous Catheters
Acronym: CAS-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Kander (Other)
Responsible Party: Sponsor-Investigator, Thomas Kander, Professor, Region Skane
Organization: Region Skane (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAS-2
Record Dates: First submitted 2025-05-12; First posted 2025-06-11 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Central Venous Catheter; Coagulation; Coagulation Activation; Central Venous Catheter Complications
Keywords: coagulation; ROTEM; central venous catheter
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Masking Description: Assossors of routine and complementary coagulation assays are masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group A: MERITMEDICAL Careflow™ (Active Comparator): Participants will receive a MERITMEDICAL Careflow™ two-lumen 7 Fr, 150 mm, polyurethane central venous catheter (OD 2.4 mm).
  Interventions: Device: MERITMEDICAL Careflow™ Two-Lumen Central Venous Catheter
- Group B: ARROW (Active Comparator): Participants will receive an ARROW two-lumen 7 Fr, 160 mm, polyurethane central venous catheter (OD 2.5 mm).
  Interventions: Device: ARROW Two-Lumen Central Venous Catheter
- Group C: ARROWg+ard Blue Plus® (Active Comparator): Participants will receive an ARROWg+ard Blue Plus® two-lumen 8 Fr, 160 mm, polyurethane catheter (OD 2.8 mm) with chlorhexidine and silver sulfadiazine coating.
  Interventions: Device: ARROWg+ard Blue Plus® Two-Lumen Central Venous Catheter
- Group D: Multicath 2 Expert UP (Active Comparator): Participants will receive a Multicath 2 Expert UP two-lumen 7.5 Fr, 160 mm, polyurethane shaft embedded with silver ions (OD 2.5 mm).
  Interventions: Device: Multicath 2 Expert UP Two-Lumen Central Venous Catheter

INTERVENTIONS:
Device: MERITMEDICAL Careflow™ Two-Lumen Central Venous Catheter — 7 Fr, 150 mm, radio-opaque polyurethane catheter (OD 2.4 mm)
  Arms: Group A: MERITMEDICAL Careflow™
Device: ARROW Two-Lumen Central Venous Catheter — 7 Fr, 160 mm, radio-opaque polyurethane catheter (OD 2.5 mm)
  Arms: Group B: ARROW
Device: ARROWg+ard Blue Plus® Two-Lumen Central Venous Catheter — 8 Fr, 160 mm, radio-opaque polyurethane catheter with antimicrobial coating
  Arms: Group C: ARROWg+ard Blue Plus®
Device: Multicath 2 Expert UP Two-Lumen Central Venous Catheter — 7.5 Fr, 160 mm, central venous catheter (OD 2.5 mm). Polyurethane shaft embedded with silver ions.
  Arms: Group D: Multicath 2 Expert UP

SUMMARY:
A central venous catheter (CVC) is a thin plastic tube placed into one of the body's large veins, typically in the neck or near the clavicle. CVCs are crucial for administering medications, fluids, and secure blood samples. Although CVCs are an essential tool in healthcare, there are certain risks and complications associated with their use. CVCs can affect the body's coagulation system, potentially leading to the formation of blood clots at the site of the catheter. This can result in serious complications, and in some cases, increased morbidity and mortality. Despite the known risk of blood clot formation with catheter use, it is still do not fully understand why clots occur or how a newly inserted catheter affects the coagulation system.

The aim of this randomized controlled trial is to compare four different central venous catheters and their impact on the coagulation system.

Eighty eight patients ≥18 years of age, who require a CVC and agree to participate in the study will be randomly assigned to one of the four predetermined, commonly used, central venous catheters. Two blood samples will be taken from the newly inserted catheter. The first blood sample (Sample 1) will be collected within seconds after catheter insertion without pre-flushing the catheter with saline. The second blood sample (Sample 2) will be taken after the catheter has been flushed with at least 10 ml saline and the initial blood discarded. All samples will be taken from the distale lumen without any connectors. Samples 1 and 2 will then be analyzed to measure how the coagulation system is affected after contact with the inside surface of the CVC. The blood samples will also be compared between the different catheter types.

The study could provide valuable information on how the coagulation system is affected after catheter insertion. This knowledge could help improve preventive measures to reduce the risk of blood clot formation and ensure safer blood sampling for patients with venous catheters.

DETAILED DESCRIPTION:
This is a randomized controlled trial, designed to evaluate coagulation activation in response to four different commercially available central venous catheters (CVCs), all with similar internal surface areas. The study focuses on comparing changes in coagulation parameters, primarily clotting time (CT), measured using rotational thromboelastometry (ROTEM® NATEM), as well as additional ROTEM variables and standard coagulation markers.

Participants are included based on clinical need for central venous access, and are randomized using REDCap to receive one of four CVC types:

1. MERITMEDICAL Careflow™ Two-Lumen Catheter (7 Fr, 150 mm, polyurethane, OD 2.4 mm)
2. ARROW Two-Lumen Catheter (7 Fr, 160 mm, polyurethane, OD 2.5 mm)
3. ARROWg+ard Blue Plus® Two-Lumen Catheter (8 Fr, 160 mm, polyurethane, OD 2.8 mm, chlorhexidine/silver sulfadiazine coating)
4. Multicath 2 Expert UP Two-Lumen Catheter (7.5 Fr, 160 mm, polyurethane shaft embedded with silver ions, OD 2.5 mm)

Blood samples will be collected at two time points for each participant:

* Sample 1: Immediately after catheter insertion, before flushing
* Sample 2: After at least 10 ml saline flush and discard protocol

All catheters will be inserted without pre-procedural filling with saline.

Blood will be collected into Vacuette® CTAD tubes (Greiner Bio-One, Kremsmünster, Austria) containing sodium citrate, theophylline, adenosine, and dipyridamole, designed for hemostatic testing. The tubes will be inverted eight times immediately after blood collection and kept at 37°C until processing. ROTEM® analysis will be performed within 3 hours of blood collection. After the ROTEM® analysis, the remaining blood will undergo centrifugation at 4000g for 15 minutes, and 600-700 µL of plasma from each sample will be transferred into cryotubes, which will be immediately frozen and stored at -80°C for further analysis.

Laboratory and ROTEM® Analyses

ROTEM® analyses will be performed on whole blood using recalcified non-activated thromboelastometry (NATEM), in accordance with the manufacturer's instructions. Each test will be run for 60 minutes, measuring the following variables:

Clotting Time (CT) - time to initial fibrin formation Clot Formation Time (CFT) - speed of thrombus development Alpha Angle (α-angle) - kinetics of clot formation Maximum Clot Firmness (MCF) - measure of final clot strength

Routine Plasma-Based Coagulation Assays:

Prothrombin Time-International Normalized Ratio (PT-INR) Activated Partial Thromboplastin Time (aPTT)

The following coagulation markers will also be assessed:

Factor VII (FVII) and Factor XII (FXII) Thrombin-Antithrombin Complex (TAT)

ELIGIBILITY:
Inclusion Criteria

Participants must meet all of the following criteria to be included in the study:

Clinical indication for the placement of a two-lumen central venous catheter (length 150-160 mm).

Age ≥18 years. Signed informed consent.

No current use of anticoagulants or platelet inhibitors, except:

* Prophylactic low molecular weight heparin (LMWH),
* Double prophylactic dose of LMWH,
* Acetylsalicylic acid (ASA).

Exclusion Criteria

Participants meeting any of the following criteria will be excluded:

* Prothrombin complex (pK/INR) outside the normal range (0.9-1.2), if already available.
* Platelet count <50 × 10⁹/L, if already available.
* Haemoglobin < 80 g/L, if already available.
* Known coagulopathic conditions, including but not limited to:
* Activated protein C (APC) resistance,
* Hemophilia A or B,
* Vitamin K deficiency,
* Disseminated intravascular coagulation (DIC),
* Antiphospholipid syndrome,
* von Willebrand disease, Other known congenital or acquired bleeding disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in ROTEM Clotting Time (CT) (seconds) between Sample 1 and Sample 2 | Immediately after catheter insertion (Sample 1) and after flush and discard, within one hour (Sample 2)
  The primary endpoint is the difference in clotting time (CT), measured using ROTEM NATEM, between two blood samples collected from each participant. Sample 1 is collected immediately after catheter insertion, and Sample 2 is collected after a standardized flush and discard procedure. The change in CT will be compared across the four catheter groups to evaluate differences in coagulation activation.

SECONDARY OUTCOMES:
Within catheter group change in Clotting Time (CT) (seconds) between Sample 1 and Sample 2 | Immediately after catheter insertion (Sample 1) and after flush and discard, within one hour (Sample 2)
  Within-catheter group changes in CT between Sample 1 and Sample 2 will be analyzed
Change in ROTEM Clot Formation Time (CFT) (seconds) between Sample 1 and Sample 2 | Immediately after catheter insertion (Sample 1) and after flush and discard, within one hour (Sample 2)
  The within-subject differences in CFT between Sample 1 and Sample 2 will be analyzed and compared across the four catheter types. In addition within-catheter group changes in CFT between Sample 1 and Sample 2 will be analyzed
Change in ROTEM Alpha Angle (α-angle) (degrees) between Sample 1 and Sample 2 | Immediately after catheter insertion (Sample 1) and after flush and discard, within one hour (Sample 2)
  The within-subject differences in α-angle between Sample 1 and Sample 2 will be analyzed and compared across the four catheter types. In addition, within-catheter group changes in α-angle between Sample 1 and Sample 2 will be analyzed
Change in ROTEM Maximum Clot Firmness (MCF) (mm) between Sample 1 and Sample 2 | Immediately after catheter insertion (Sample 1) and after flush and discard, within one hour (Sample 2)
  The within-subject differences in MCF between Sample 1 and Sample 2 will be analyzed and compared across the four catheter types. In addition, within-catheter group changes in MCF between Sample 1 and Sample 2 will be analyzed
Change in Prothrombin Time - International Normalized Ratio (PT-INR) (continous unitless variable) between Sample 1 and Sample 2 | Immediately after catheter insertion (Sample 1) and after flush and discard, within one hour (Sample 2)
  The within-subject differences in PT-INR between Sample 1 and Sample 2 will be analyzed and compared across the four catheter types. In addition, within-catheter group changes in PT-INR between Sample 1 and Sample 2 will be analyzed
Change in Activated Partial Thromboplastin Time (aPTT) (seconds) between Sample 1 and Sample 2 | Immediately after catheter insertion (Sample 1) and after flush and discard, within one hour (Sample 2)
  The within-subject differences in aPTT between Sample 1 and Sample 2 will be analyzed and compared across the four catheter types. In addition, within-catheter group changes in aPTT between Sample 1 and Sample 2 will be analyzed
Change in Factor VII Activity (FVII) (kIU/L) between Sample 1 and Sample 2 | Immediately after catheter insertion (Sample 1) and after flush and discard, within one hour (Sample 2)
  The within-subject differences in FVII between Sample 1 and Sample 2 will be analyzed and compared across the four catheter types. In addition, within-catheter group changes in FVII between Sample 1 and Sample 2 will be analyzed
Change in Factor XII Activity (FXII) (kIU/L) between Sample 1 and Sample 2 | Time Immediately after catheter insertion (Sample 1) and after flush and discard, within one hour (Sample 2)
  The within-subject differences in FXII between Sample 1 and Sample 2 will be analyzed and compared across the four catheter types. In addition, within-catheter group changes in FXII between Sample 1 and Sample 2 will be analyzed
Change in Thrombin-Antithrombin Complex Concentration (TAT) (mikrogr/L) between Sample 1 and Sample 2 | Immediately after catheter insertion (Sample 1) and after flush and discard, within one hour (Sample 2)
  The within-subject differences in TAT between Sample 1 and Sample 2 will be analyzed and compared across the four catheter types. In addition, within-catheter group changes in TAT between Sample 1 and Sample 2 will be analyzed

CONTACTS AND LOCATIONS:
Locations (1):
- Skåne University Hospital Lund, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the study results will be made available upon reasonable request. Data will be completely anonymized prior to sharing, in accordance with applicable data protection regulations. Requests from both academic researchers and commercial entities (e.g., device manufacturers) will be considered. All requests will undergo review to assess scientific validity and compliance with ethical standards.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available starting 6 months after publication of the primary results and will remain available for 5 years.
Access Criteria: Access will be granted to researchers or organizations submitting a methodologically sound proposal. Approval is at the discretion of the study investigators, subject to compliance with applicable regulations and ethical considerations.

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-08-29): https://cdn.clinicaltrials.gov/large-docs/22/NCT07014722/SAP_000.pdf